CLINICAL TRIAL: NCT00534248
Title: A Phase III Clinical Trial to Evaluate the Efficacy, Immunogenicity, Safety and Tolerability of Zostavax™ in Subjects 50-59 Years of Age
Brief Title: Study to Evaluate the Safety and Effectiveness of Zostavax™ in Subjects 50 - 59 Years of Age (V211-022)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V211-022; 2007_551
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Results first posted 2011-05-02 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Shingles
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Zostavax™ (Experimental): Participants randomized to receive Zoster Vaccine, Live (Zostavax™).
  Interventions: Biological: Zoster Vaccine, Live (Zostavax™)
- Placebo (Placebo Comparator): Participants randomized to receive Placebo.
  Interventions: Biological: Comparator: Placebo

INTERVENTIONS:
Biological: Zoster Vaccine, Live (Zostavax™) — A single dose 0.65 ml Zostavax™ (Live, attenuated Zoster Vaccine) was administered by subcutaneous injection on Day 1.
  Other Names: V211; Zostavax™
  Arms: Zostavax™
Biological: Comparator: Placebo — A single dose of 0.65 ml Placebo (A vaccine stabilizer of Zostavax™ with no live virus) was administered by subcutaneous injection on Day 1.
  Arms: Placebo

SUMMARY:
This study will look at how well Zostavax™ works in preventing shingles in participants ages 50-59 years old.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 50 - 59 years of age
* No fever on day of vaccination
* Females of reproductive potential must be willing to use acceptable form of birth control

Exclusion Criteria:

* Have received chicken pox or shingles vaccine
* Have already had shingles
* Have recently had another vaccination
* Pregnant or breast feeding. Have participated in another research study in the last 30 days
* You are taking certain antiviral drugs
* History of allergic reaction to any vaccine component, including gelatin or neomycin

Ages: 50 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22439 (Actual)
Dates: Start 2007-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Gilbert PB, Gabriel EE, Miao X, Li X, Su SC, Parrino J, Chan IS. Fold rise in antibody titers by measured by glycoprotein-based enzyme-linked immunosorbent assay is an excellent correlate of protection for a herpes zoster vaccine, demonstrated via the vaccine efficacy curve. J Infect Dis. 2014 Nov 15;210(10):1573-81. doi: 10.1093/infdis/jiu279. Epub 2014 May 13. PMID 24823623
- [Derived] Levin MJ, Schmader KE, Gnann JW, McNeil SA, Vesikari T, Betts RF, Keay S, Stek JE, Bundick ND, Su SC, Zhao Y, Li X, Chan IS, Annunziato PW, Parrino J. Varicella-zoster virus-specific antibody responses in 50-59-year-old recipients of zoster vaccine. J Infect Dis. 2013 Nov 1;208(9):1386-90. doi: 10.1093/infdis/jit342. Epub 2013 Aug 1. PMID 23908486
- [Derived] Schmader KE, Levin MJ, Gnann JW Jr, McNeil SA, Vesikari T, Betts RF, Keay S, Stek JE, Bundick ND, Su SC, Zhao Y, Li X, Chan IS, Annunziato PW, Parrino J. Efficacy, safety, and tolerability of herpes zoster vaccine in persons aged 50-59 years. Clin Infect Dis. 2012 Apr;54(7):922-8. doi: 10.1093/cid/cir970. Epub 2012 Jan 30. PMID 22291101

RESULTS

PARTICIPANT FLOW:
Groups:
- Zostavax™: Participants randomized to receive a single 0.65 ml subcutaneous injection of Zoster Vaccine, Live (Zostavax™).
- Placebo: Participants randomized to receive a single 0.65 ml subcutaneous injection of placebo.
Period: Overall Study
Arm/Group | Zostavax™ | Placebo
Started | 11211 | 11228
VACCINATED | 11186 | 11210
Completed | 10550 | 10555
Not Completed | 661 | 673
Not completed — Adverse Event | 19 | 29
Not completed — Lost to Follow-up | 353 | 375
Not completed — Other protocol specified criteria | 13 | 3
Not completed — Physician Decision | 10 | 7
Not completed — Protocol Violation | 3 | 4
Not completed — Withdrawal by Subject | 263 | 255

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zostavax™ | Placebo | Total
Number analyzed (Participants) | 11211 | 11228 | 22439
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (2.8) | 54.8 (2.8) | 54.8 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6913 | 6972 | 13885
  Male | 4298 | 4256 | 8554

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Confirmed Herpes Zoster (HZ) Cases by Vaccination Group
Description: Incidence rate of HZ cases was defined as the number of confirmed HZ cases per 1000 person-years of follow-up following vaccination. Vaccine efficacy for HZ was defined as the relative reduction in incidence rate of HZ in the group that received Zostavax™ compared with the group that received placebo based on the intent-to-treat population.
Time Frame: 2 Years
Population: Intent-to-treat population defined as all participants randomized in the study according to the planned treatment, Zostavax or placebo, they were assigned.
Measure: Mean (95% Confidence Interval); unit: number of HZ cases/1000 person-years
Arm/Group | Zostavax™ | Placebo
Number analyzed (Participants) | 11211 | 11228
number of HZ cases/1000 person-years | 1.994 [1.346 to 2.847] | 6.596 [5.361 to 8.030]
Statistical Analysis 1: Comparison: Zostavax™ vs Placebo; Vaccine efficacy with respect to HZ was defined as the relative reduction in incidence rate of HZ point estimate (95% CI) calculated as 1 minus the ratio of the estimated incidence rates of HZ in the zoster vaccine group and the placebo group; Test type: Superiority or Other; p < .001, Conditional Exact Method; point estimate = .698, 95% CI 2-sided [.541 to .806] — The point estimate was for vaccine efficacy with respect to incidence of HZ

2. Secondary Outcome: Varicella-zoster Virus (VZV) Antibody Response at 6 Weeks Post Vaccination by Vaccination Group
Description: VZV antibody response as measured by Glycoprotein Enzyme-Linked Immunosorbent Assay (gpELISA) in the group that received Zostavax™ compared with the group that received placebo, based on the random subcohort population.
Time Frame: 6 Weeks
Population: Random subcohort population included 10% of all randomized participants randomly selected for immunogenicity assay, were vaccinated (according to actual treatment received), had results at prevaccination and at 6 weeks postvaccination. Results from participants with protocol violations that may impact the immunogenicity analysis were excluded.
Measure: Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | Zostavax™ | Placebo
Number analyzed (Participants) | 1088 | 1087
gpELISA units/mL | 660.0 [624.7 to 697.2] | 293.1 [274.7 to 312.6]
Statistical Analysis 1: Comparison: Zostavax™ vs Placebo; Test type: Superiority or Other; p < .001, linear mixed longitudinal analysis model; geometric mean titre ratio = 2.3, 95% CI 2-sided [2.2 to 2.4]

3. Secondary Outcome: Number of Participants Reporting One or More Serious Adverse Experiences by Vaccination Group During the 42-day Postvaccination Follow-up Period
Description: A serious adverse event is defined as any adverse event that results in death, is life threatening, results in a persistent or significant disability/incapacity, results in hospitalization or prolongs an existing
  hospitalization, is a congenital anomaly/birth defect, is a cancer, is an overdose, or is considered an "other important medical event" based on medical judgement.
Time Frame: Through 42 days post-vaccination
Population: All participants who were vaccinated according to actual treatment received (Zostavax or placebo) and had safety follow-up.
Measure: Number; unit: participants
Arm/Group | Zostavax™ | Placebo
Number analyzed (Participants) | 11094 | 11116
participants | 69 [.48 to .79] | 61 [.42 to .70]
Statistical Analysis 1: Comparison: Zostavax™ vs Placebo; Analysis of proportion of participants reporting one or more serious adverse experiences reported within 42 days postvaccination; Test type: Superiority or Other; Relative Risk = 1.133, 95% CI 2-sided [.805 to 1.595]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) are presented that occurred from Day 1 to 182 postvaccination. Deaths that occurred any time during the study are also included. Non-serious AEs are presented for events that occurred from Day 1 to 42 postvaccination.
Description: AEs and SAEs were reported in participants who were vaccinated according to actual treatment received (Zostavax or placebo) and had safety follow-up.
Arm/Group | Zostavax™ | Placebo
Serious Adverse Events (participants affected / at risk) | 243/11094 | 233/11116
Other Adverse Events (participants affected / at risk) | 7228/11094 | 2183/11116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zostavax™ (N=11094) | Placebo (N=11116)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 6 (6)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 5 (5) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 2 (2)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (4) | 5 (5)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Congenital diaphragmatic hernia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Porphyria acute (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatic disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 7 (7) | 7 (7)
Death (General disorders) | 3 (3) | 2 (2)
Hernia obstructive (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 5 (5) | 7 (7)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Perforation bile duct (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic oedema (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 6 (6) | 7 (7)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bursitis infective staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 5 (5)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diabetic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (3) | 2 (2)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Epidemic nephropathy (Infections and infestations) | 2 (2) | 1 (1)
Erysipelas (Infections and infestations) | 4 (4) | 2 (2)
Furuncle (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 8 (8)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Bladder injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Device failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stent occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ureteric injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 10 (10)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of cervix uteri (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 7 (7)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 3 (3)
Cervical root pain (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Facial palsy (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 2 (2) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 3 (6)
Completed suicide (Psychiatric disorders) | 0 (0) | 3 (3)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 1 (1)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Drug dependence (Psychiatric disorders) | 1 (2) | 0 (0)
Major depression (Psychiatric disorders) | 2 (2) | 2 (2)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zostavax™ (N=11094) | Placebo (N=11116)
Injection site erythema (General disorders) | 5351 (5409) | 483 (484)
Injection site pain (General disorders) | 6005 (6276) | 1025 (1052)
Injection site pruritus (General disorders) | 1287 (1307) | 78 (84)
Injection site swelling (General disorders) | 4500 (4549) | 309 (311)
Headache (Nervous system disorders) | 1041 (1509) | 917 (1357)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less